CLINICAL TRIAL: NCT06196203
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase 2 Study of AK117/Placebo in Combination With Azacitidine in Patients With Newly Diagnosed Higher-risk Myelodysplastic Syndromes
Brief Title: A Study of AK117 in Combination With Azacitidine in Patients With Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK117-205
Record Dates: First submitted 2023-12-24; First posted 2024-01-09 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Higher-risk Myelodysplastic Syndromes
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AK117 (dose 1) in combination with azacitidine (Experimental): Subjects receive AK117 (dose 1) intravenously, in combination with azacitidine (75 mg/m2, D1-7, Q4W) subcutaneously
  Interventions: Drug: AK117; Drug: Azacitidine
- AK117 (dose 2) in combination with azacitidine (Experimental): Subjects receive AK117 (dose 2) intravenously, in combination with azacitidine (75 mg/m2, D1-7, Q4W) subcutaneously
  Interventions: Drug: AK117; Drug: Azacitidine
- Placebo in combination with azacitidine (Placebo Comparator): Subjects receive placebo intravenously, in combination with azacitidine (75 mg/m2, D1-7, Q4W) subcutaneously
  Interventions: Drug: Placebo; Drug: Azacitidine

INTERVENTIONS:
Drug: AK117 — AK117 IV injection
  Arms: AK117 (dose 1) in combination with azacitidine; AK117 (dose 2) in combination with azacitidine
Drug: Placebo — Placebo IV injection
  Arms: Placebo in combination with azacitidine
Drug: Azacitidine — Azacitidine SC injection

SUMMARY:
This is a Phase 2 randomized, double-blind, placebo-controlled, multicenter study evaluating the efficacy and safety of AK117 or placebo, combined with azacitidine in patients with newly diagnosed higher-risk myelodysplastic syndromes (HR-MDS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of enrolment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2.
* Expected life expectancy ≥ 3 months.
* Newly diagnosed HR-MDS, according to the 2016 World Health Organization (WHO) classification with the presence of < 20% blasts in bone marrow or peripheral blood; Overall IPSS-R score ≥ 3.5.
* Ability to undergo the study-required bone marrow sample collection procedures.
* Suitable venous access for the study-required blood sampling (i.e., including PK and immunogenicity).
* Female patients of childbearing age must have negative serum pregnancy test results before randomization or per region-specific guidance documented in the informed consent and a negative urine pregnancy test on the day of first dose prior to dosing.
* Female patients of childbearing potential having sex with an unsterilized male partner must agree to use a highly effective method of contraception from the beginning of screening until 180 days after the last dose of the study treatment.
* Unsterilized male patients having sex with a female partner of childbearing potential must agree to use an effective method of contraception from the beginning of screening until 180 days after the last dose of study treatment.

Exclusion Criteria:

* MDS evolving from a pre-existing myeloproliferative neoplasm (MPN), myelodysplastic/myeloproliferative neoplasms (MDS/MPN).
* Prior treatment with Cluster of Differentiation (CD) 47 or Signal-regulatory protein alpha (SIRPα)-targeting agents.
* Concurrently participating in another interventional clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Patients who previously diagnosed with another malignancy and have any evidence of residual disease.
* Known allergy to any component of any study drug; known history of severe hypersensitivity to other monoclonal antibodies.
* Patients with any psychiatric or social factor which the investigator deems may interfere with the patient's ability to comply with the requirements of the study.
* Patients with current hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy.
* Patients with known cardiopulmonary disease defined as unstable angina, clinically significant arrhythmia, congestive heart failure (New York Heart Association Class III or IV), decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders.
* Patients who are breastfeeding or plans to breastfeed during the study.
* Other conditions where the investigator considers the patient inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CRR) | Up to approximately 2 years
  CRR is defined as the proportion of subjects with complete remission (CR) per International Working Group (IWG) 2023 criteria

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 2 years
  The proportion of subjects with recorded response per IWG 2023
Time to response (TTR) | Up to approximately 2 years
  Time from the randomization to the first recorded response
Time to CR (TTCR) | Up to approximately 2 years
  Time from the randomization to the first recorded CR
Duration of response (DoR) | Up to approximately 2 years
  Time from the first recorded response until disease relapse or progression or death due to any cause, whichever occurs first
Duration of CR (DoCR) | Up to approximately 2 years
  Time from the first recorded CR until disease relapse or progression or death due to any cause, whichever occurs first
Event-free survival (EFS) | Up to approximately 2 years
  Time from randomization until transformation to AML or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 2 years
  The time from randomization until death due to any cause
Number of subjects with adverse events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Pharmacokinetic characteristics | Up to approximately 2 years
  Serum concentrations of AK117 in individual subjects at different time points after AK117 administration
Anti-drug antibody (ADA) | Up to approximately 2 years
  Number of subjects with detectable anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - American Oncology Partners, PA (The Center for Cancer and Blood Disorders-Bethesda), Bethesda, Maryland
  - Maryland Oncology-Columbia, Columbia, Maryland
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
- Institute of hematolongy&blood diseases hospital, chinese academy of medical sciences&peking union medical college, Tianjin, China

IPD SHARING:
Plan to Share IPD: No